CLINICAL TRIAL: NCT02451163
Title: A Randomized, Controlled Clinical Study on the Effect of Polysaccharides From Wheat on Common Cold Infections in Elderly
Brief Title: DBRCT on the Effect of Wheat Polysaccharides on Common Cold Infections in Elderly
Acronym: Fib-CC-2014
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clinical Research Center Kiel GmbH (Other)
Collaborators: BioActor (Industry); European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Fib-CC-2014
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Upper Respiratory Infections; Common Cold
MeSH Terms: conditions — Respiratory Tract Infections; Common Cold | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- polysaccharides from wheat (Active Comparator): 12.0 g powder containing 10.0 g active ingredient (wheat polysaccharides) as well as 2.0 g filling substance (maltodextrin) stirred in milk or filtered apple juice (200 ml each).
  Interventions: Dietary Supplement: wheat polysaccharides
- control product (Placebo Comparator): 12.0 g maltodextrin stirred in milk or filtered apple juice (200 ml each).
  Interventions: Dietary Supplement: maltodextrin

INTERVENTIONS:
Dietary Supplement: wheat polysaccharides — Consumed once daily for 12 weeks.
  Arms: polysaccharides from wheat
Dietary Supplement: maltodextrin — Consumed once daily for 12 weeks.
  Arms: control product

SUMMARY:
The aim of the study is to measure the effect of wheat polysaccharides on the occurence of common cold (CC) in elderly during a 12-week consumption period.

DETAILED DESCRIPTION:
The study is conducted in the frame of the collaborative project 'FibeBiotics' (No. 289517) (Fibers as support of the Gut and Immune function of Elderly - From polysaccharide compound to health Claim) within the Seventh Framework Programme (FP7) for Research and Technological Development of the European Union (EU).

ELIGIBILITY:
Inclusion Criteria:

* men and postmenopausal women aged ≥ 50
* willingness to abstain as far as possible from food and supplements containing probiotics, prebiotic supplements, other fermented products, supplements containing vitamins and minerals as well as willingness to sustain a low dietary fibre diet for 14 weeks
* written informed consent

Exclusion Criteria:

* subjects currently enrolled in another clinical study
* subjects having finished another clinical study within the last 4 weeks before inclusion
* surgery or intervention requiring general anaesthesia within 2 months before the study
* current symptoms of common infectious diseases (CID) of the airways or other organ systems e.g. gastrointestinal tract
* history of allergic rhinitis, allergic asthma, anaphylactic shock, quincke edema, food allergy (type I allergy)
* allergy or hypersensitivity to any component of the test product (e. g. wheat, corn)
* known congenital, acquired or iatrogenic immunodeficiency (e.g. HIV, chemotherapy, immunosuppression)
* active autoimmune diseases
* severe chronic disease (COPD, respiratory insufficiency, cancer, IBD, malabsorption, malnutrition, chronic inflammatory diseases, severe renal, hepatic or cardiac diseases)
* known coeliac disease (gluten enteropathy)
* chronic systemic or chronic topical treatment likely to interfere with evaluation of the study parameters: antiallergic drugs, antibiotics, intestinal or respiratory antiseptics, anti-rheumatics, antiphlogistics (except aspirin or equivalent products preventing from aggregation of platelets or blood clotting) and steroids prescribed in chronic inflammatory diseases (in the last 4 weeks before inclusion)
* diabetes mellitus
* other chronic treatments likely to interfere with study outcome: e.g. laxatives, body weight management and/or medication
* chronic abdominal pain
* bowel movement less than 3 times per week
* subjects, who meet 2 or more Rome III criteria for constipation or who take laxatives on a regular basis
* vegetarian, vegan diet
* eating disorders (e.g. anorexia, bulimia)
* alcohol and drug abuse
* severe neurological, cognitive or psychiatric diseases
* subjects not understanding or speaking fluently German
* legal incapacity

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Occurrence of common cold (CC) based on Jackson et al. 1958 and physicians diagnosis | 12 weeks
  Occurrence of common cold (= number of subjects affected by at least one common cold episode during intervention) according to self-reporting (questionnaire based on Jackson et al. 1958) and physicians diagnosis.

SECONDARY OUTCOMES:
Cumulative severity of common cold episodes | 12 weeks
  Cumulative severity of common cold episodes (= sum of daily symptom scores acc. to Jackson et al. 1958).

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Laue, MD, Principal Investigator — Clinical Research Center Kiel GmbH
Locations (1):
- Clinical Research Center (CRC) Kiel GmbH, Kiel, Schleswig-Holstein, Germany